CLINICAL TRIAL: NCT06837584
Title: A Multicenter Observational Study on the Current Status of Control and Treatment of Outpatient Children With Asthma and the Types of Airway Inflammation
Brief Title: Control and Treatment of Outpatient Children With Asthma
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Kunling Shen, Professior, Shenzhen Children's Hospital
Other Study IDs: Asthma 002
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Asthma
Keywords: asthma; children; outpatients; management; control
MeSH Terms: conditions — Asthma | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Questionnaire and Physical Exam

SUMMARY:
The aim of this study is to comprehensively understand the disease control and management status of children with asthma in China, as well as the types of airway inflammation. The findings of this survey will help improve the asthma control level in Chinese children, facilitate future patient education, and guide rational medication use. Moreover, it will provide important evidence for health decision-making departments to better allocate and utilize medical resources.

DETAILED DESCRIPTION:
Bronchial asthma (hereinafter referred to as asthma) is the most common chronic respiratory disease in children. It severely affects the physical and mental health of children and imposes a huge economic burden on families and society, consuming a large amount of medical and health resources. In recent years, the prevalence of asthma in children worldwide has generally continued to rise. Data from the Global Burden of Disease database in 2019 showed that the prevalence of asthma in children aged 0-9 years was 4.21%, in children aged 10-14 years was 4.10%, and in adolescents aged 15-19 years was 3.00%. In China, over the past 20 years, the prevalence of asthma in children has also shown an overall upward trend, increasing from 0.91% in 1990 to 1.54% in 2000, and then to 3.02% in 2010. Thanks to the continuous efforts of several generations of pediatricians, the level of standardized diagnosis and treatment of childhood asthma has significantly improved. However, the control of asthma in children still faces many challenges.

The purpose of this study is to comprehensively understand the disease control and management status of children with asthma in China, as well as the types of airway inflammation. The findings of this survey will help improve the asthma control level in Chinese children, facilitate future patient education, guide rational medication use, and provide important evidence for health decision-making departments to better allocate and utilize medical resources.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 and 18 years old
* Diagnosed with asthma for more than 3 months
* Had asthma symptoms or asthma treatment within the past 12 months.

Exclusion Criteria:

* With other respiratory diseases such as bronchiectasis, bronchiolitis, cystic fibrosis, and pneumonia
* Have participated in any interventional clinical studies related to asthma within the 3 months prior to enrollment in this study
* Parents, legal representatives, or guardians do not agree to participate in this study.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 2-16 years and diagnosed with asthma ≥3 months were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 42000 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Asthma control level | 3 months before and at the time of enrollment
  The Asthma Control Test (ACT) will be employed for assessment, with the following interpretation criteria: a total score of 20-25 indicates well-controlled asthma, where symptoms are satisfactorily managed and the current treatment regimen should be continued; a score of 16-19 suggests poorly controlled asthma, indicating suboptimal symptom management that requires treatment adjustment or enhanced disease management; and a score of 5-15 reflects very poorly controlled asthma, with severe uncontrolled symptoms necessitating immediate medical attention and treatment modification.
The proportion of type 2 inflammation | 3 months before and at the time of enrollment
  Blood EOS and IgE were used to judge. The T2 inflammatory phenotypes were classified based on blood eosinophil count and total specific IgE levels: Only-atopy was defined as blood eosinophils <300/μL with sum of all specific IgE ≥0.7 kU/L; Only-EOS as blood eosinophils ≥300/μL with sum of all specific IgE <0.7 kU/L; T2-high as blood eosinophils ≥300/μL with sum of all specific IgE ≥0.7 kU/L; and T2-low as blood eosinophils <300/μL with sum of all specific IgE <0.7 kU/L.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol